CLINICAL TRIAL: NCT07074457
Title: A Prospective, Exploratory Clinical Study of Chidamide Combined With Brentuximab Vedotin Regimen in the Treatment of CD30 Positive PTCL Patients Unfit for Chemotherapy
Brief Title: Chidamide Combined With Brentuximab Vedotin Regimen for CD30+ PTCL Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024470
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: CD30+ Peripheral T-cell Lymphoma
Keywords: Chidamide; Brentuximab vedotin; Unfit for chemotherapy
MeSH Terms: interventions — Brentuximab Vedotin; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (patients achieved CR) (Experimental): Patients achieving CR after 3 cycles of BvC therapy will receive 3 additional cycles of BvC consolidation followed by chidamide maintenance therapy for ≥2 years
  Interventions: Drug: Induction therapy-3 cycles of BvC (Brentuximab vedotin plus Chidamide); Drug: Consolidation therapy- 3 or 6 cycles of BvC(Brentuximab vedotin plus chidamide); Drug: Maintenance therapy-chidamide
- Cohort 2 (patients achieved PR) (Experimental): Patients achieving PR after 3 cycles of BvC therapy will receive 6 additional cycles of BvC consolidation followed by chidamide maintenance therapy for ≥2 years
  Interventions: Drug: Induction therapy-3 cycles of BvC (Brentuximab vedotin plus Chidamide); Drug: Consolidation therapy- 3 or 6 cycles of BvC(Brentuximab vedotin plus chidamide); Drug: Maintenance therapy-chidamide

INTERVENTIONS:
Drug: Induction therapy-3 cycles of BvC (Brentuximab vedotin plus Chidamide) — 3 cycles of BvC treatment for all enrolled patients.
  Brentuximab vedotin; Specification: 50mg per vial; 1.8mg/kg qd d1 every 3 weeks, ivgtt.;
  Chidamide; Specification: 5mg per tablet; 20mg biw for 2 weeks every 3 weeks, po.;
Drug: Consolidation therapy- 3 or 6 cycles of BvC(Brentuximab vedotin plus chidamide) — Consolidation therapy( For patients who achieved CR after induction therapy, 3 cycles of additional BvC treatment; For patients who achieved PR after induction therapy, 6 cycles of additional BvC treatment).
  Brentuximab vedotin; Specification: 50mg per vial; 1.8mg/kg qd d1 every 3 weeks, ivgtt.;
  Chidamide; Specification: 5mg per tablet; 20mg biw for 2 weeks every 3 weeks, po.;
  Maintenance therapy chidamide (20mg biw for 2 weeks every 3 weeks, po.) for ≥2 years
Drug: Maintenance therapy-chidamide — Chidamide (20mg biw for 2 weeks every 3 weeks, po.) for ≥2 years

SUMMARY:
To evaluate the efficacy and safety of chidamide combined with brentuximab vedotin regimen for CD30 positive PTCL patients who are unfit for chemotherapy.

DETAILED DESCRIPTION:
This study will enroll CD30-positive peripheral T-cell lymphoma (PTCL) patients who are ineligible for conventional chemotherapy. Participants will receive induction therapy with 3 cycles of BvC regimen (brentuximab vedotin plus chidamide combination). Patients demonstrating disease progression (PD) or stable disease (SD) will be withdrawn from the study. Patients achieving partial remission(PR) or complete remission(CR) will receive stratification consolidation therapy as followings:

Cohort 1 (patients achieved CR): Receive 3 additional cycles of BvC consolidation

Cohort 2 (patients achieved PR): Receive 6 additional cycles of BvC consolidation

After consolidation therapy, responding patients (CR/PR) will receive chidamide maintenance therapy for ≥2 years

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥70 years or age < 70 years and unfit for chemotherapy, male or female not limited;
2. Patients must have the capacity to understand and willingly provide written informed consent;
3. ECOG score 0-3 points;
4. Expected lifespan>3 months;
5. Patients with CD30+ peripheral T-cell lymphoma (PTCL) confirmed by histopathology/cytology using the 2022 World Health Organization (WHO) Classification of Diseases;
6. Measurable lesions with a short diameter of ≥15mm defined by PET/CT.
7. R/R PTCL: patients with at least previous first-line treatment failure and no prior exposure to chidamide and brentuximab vedotin.
8. Patients are unfit for chemotherapy after evaluation or are not considered for chemotherapy for other reasons;
9. Any non-hematological toxicity, except hair loss, associated with prior treatment in patients with R/R disease, as per NCI CTCAE version 5.0, must be managed and resolved to at least grade 1;
10. Appropriate organ function: Cardiac function: ejection fraction ≥ 50%, asymptomatic arrhythmia; Liver function: alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal, total bilirubin<2 times the upper limit of normal; Renal function: serum creatinine clearance rate ≥ 80 mL/min, creatinine<160 umol/l; Pulmonary function: Without oxygen inhalation, SPO2>90%, FEV1, FVC, and DLCO ≥ 50% predicted values;
11. Adequate bone marrow reserve is defined as: Hemoglobin ≥ 9g/dL, Platelet count ≥ 70 × 10 ^ 9/L, The absolute value of neutrophils is ≥ 1.0 × 10 ^ 9/L, If accompanied by bone marrow invasion, platelet count ≥ 50 × 10 ^ 9/L, absolute neutrophil count ≥ 0.75 × 10 ^ 9/L, The number of CD34+cells is ≥ 2.0 × 109/kg;
12. Subjects with fertility or potential for fertility must be willing to undergo contraception from the date of registration in this study until the study follow-up period;
13. Patients with good compliance.

Exclusion Criteria:

1. Patients with R/R disease previously used chidamide and brentuximab vedotin or received any other anti-tumor therapy within 4 weeks.
2. Patients enrolled in another clinical study within 4 weeks;
3. HIV infection and/or active hepatitis B or C;
4. Uncontrolled active infections;
5. Severe liver and kidney dysfunction (alanine aminotransferase, bilirubin, creatinine>3 times the upper limit of normal);
6. Existence of organic heart disease or severe arrhythmia, leading to clinical symptoms or abnormal heart function (NYHA functional class ≥ 2);
7. Simultaneously present other tumors that require treatment or intervention;
8. Previous or current history of vascular embolism;
9. Pregnant or lactating women;
10. In a state of severe immune suppression;
11. Other psychological conditions that hinder patients from participating in research or signing informed consent forms.
12. Patients are unlikely to complete all protocol study visits and procedures or do not meet the requirements for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate(CRR) | At the end of 3 cycles of BvC (each cycle is 21 days)
  The rate of patients who achieved CR after 3 cycles of BvC regimen

SECONDARY OUTCOMES:
Main adverse reactions | From enrollment to 1 month after consolidation treatment of the last patient
  The safety and tolerability of the therapeutic regimen measured by the major adverse events.
2-year overall survival(OS) | From enrollment to 2 year after treatment of the last patient
  OS will be assessed from the start of the combination regimen to the date of death or end of follow-up.
Overall response rate(ORR) | At the end of 3 cycles of BvC (each cycle is 21 days)
  The rate of patients who achieved CR or PR after 3 cycles of BvC regimen
2-year progression-free survival(PFS) | From enrollment to 2 year after treatment of the last patient
  PFS will be assessed from the first drug given to the date of progression, relapse, death or end of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China